CLINICAL TRIAL: NCT07220694
Title: An 8-week Study Evaluating the Effects of a Dietary Supplement (Sabroxy®) on Insulin Resistance and Cognitive Function in Subjects With Mild Cognitive Impairment and Insulin Resistance
Brief Title: Effects of Sabroxy® Supplementation on Insulin Resistance and Cognitive Function in Adults With Mild Cognitive Impairment and Insulin Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Sabinsa Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB20251021- A
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance; Mild Cognitive Impairment; Cognitive Decline; Neurodegenerative Disorders
Keywords: BioPerine; Insulin Sensitivity; Cognitive Function; Memory Performance; Sabroxy
MeSH Terms: conditions — Insulin Resistance; Cognitive Dysfunction; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (Sabroxy®) (Active Comparator): Subjects are to take two capsules with water in the am.
  Interventions: Dietary Supplement: Sabroxy®
- Placebo (Inactive capsule) (Placebo Comparator): Subjects are to take two capsules with water in the am.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sabroxy® — Sabroxy® is a standardized extract of Oroxylum indicum bark formulated with BioPerine® (black pepper extract) to enhance bioavailability. Each capsule contains 250 mg of Sabroxy® and 5 mg of BioPerine®, administered once daily after breakfast with water for 8 weeks.
  Sabroxy® is standardized for bioactive flavonoids such as oroxylin A, baicalein, and chrysin, which are known for their antioxidant, neuroprotective, and anti-inflammatory properties.
  The product will be supplied by Sabinsa Corporation (East Windsor, NJ, USA) under Good Manufacturing Practice (GMP) conditions and will be packaged in identical capsules to maintain blinding.
  The intervention aims to evaluate the effects of Sabroxy® on insulin resistance, inflammation, and cognitive performance in adults with mild cognitive impairment and insulin resistance.
  Other Names: Oroxylum indicum bark extract, Sabroxy® 250 mg + BioPerine® 5 mg
  Arms: Dietary Supplement (Sabroxy®)
Other: Placebo — The placebo consists of identical capsules containing inert excipients (microcrystalline cellulose and magnesium stearate) with no active botanical ingredients.
  The capsules are identical in appearance, weight, color, and packaging to the Sabroxy® capsules to maintain blinding.
  Participants assigned to the placebo group will receive one capsule orally once daily after breakfast with water for 8 weeks.
  The placebo will be manufactured and supplied under Good Manufacturing Practice (GMP) conditions by Sabinsa Corporation (East Windsor, NJ, USA).
  This control group will enable comparison of Sabroxy®'s efficacy and safety against a non-active formulation to validate clinical outcomes.
  Other Names: Matching Placebo Capsule
  Arms: Placebo (Inactive capsule)

SUMMARY:
This randomized, double-blind, placebo-controlled, 8-week clinical trial is designed to evaluate the effects of Sabroxy®, a standardized extract of Oroxylum indicum bark, on insulin resistance and cognitive function in adults with mild cognitive impairment and insulin resistance.

A total of 120 participants (men and women, aged 40-80 years) who are non-smokers, with fasting glucose levels between 100-135 mg/dL, HOMA-IR value ≥ 2.0 to < 4.0, and a Montreal Cognitive Assessment (MoCA) score below 26, will be enrolled. Eligible participants will be randomized (1:1) to receive either Sabroxy® (250 mg with 5 mg BioPerine®) or placebo, administered orally once daily for 8 weeks.

The primary endpoint is the change in insulin resistance from baseline to Week 8, assessed using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR).

The secondary endpoints include changes in:

Cognitive performance, assessed using the Immediate Word Recall, Numeric Working Memory, Cognitive Failures Questionnaire (CFQ), and Montreal Cognitive Assessment (MoCA).

Biomarkers of metabolic and neuronal function, including Brain-Derived Neurotrophic Factor (BDNF), high-sensitivity C-reactive protein (hs-CRP), fasting insulin, fasting glucose, and phosphorylated tau/amyloid beta (p-Tau/Aβ) ratio.

Safety will be assessed through adverse event monitoring, vital signs, and routine clinical laboratory tests.

The study will be conducted at a single site, San Francisco Research Institute (USA), in compliance with the Declaration of Helsinki, ICH-GCP guidelines, and 21 CFR Part 312 (where applicable).

This study seeks to generate clinical evidence supporting the potential of Sabroxy® supplementation to improve glucose tolerance, reduce inflammation, and enhance cognitive function in individuals with early metabolic and neurocognitive dysfunctions.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) often occurs alongside metabolic disturbances such as insulin resistance and chronic inflammation, which are recognized contributors to neurodegenerative risk. Sabroxy® is a standardized extract of Oroxylum indicum bark, traditionally used in Ayurvedic medicine, and has demonstrated antioxidant, neuroprotective, and glucose-regulatory properties in preclinical studies.

This study aims to evaluate the potential of Sabroxy® supplementation to improve both metabolic and cognitive outcomes in adults with MCI and insulin resistance. The trial follows a randomized, double-blind, placebo-controlled design, with 120 eligible participants randomized in a 1:1 ratio to receive either Sabroxy® (250 mg combined with 5 mg BioPerine®) or placebo once daily for 8 weeks.

The primary objective is to assess the effect of Sabroxy® on insulin resistance as measured by HOMA-IR. Secondary objectives include assessing cognitive function improvements (using Immediate Word Recall, Numeric Working Memory, CFQ, and MoCA tests), as well as evaluating changes in biochemical markers related to neuronal health (BDNF, p-Tau/Aβ ratio) and inflammation (hs-CRP).

Safety assessments include adverse event monitoring, vital signs, and standard clinical laboratory evaluations throughout the study. All study procedures are conducted at the San Francisco Research Institute (USA) in accordance with the Declaration of Helsinki, ICH-GCP guidelines, and 21 CFR Part 312 (where applicable).

The outcomes from this study are expected to contribute evidence on the dual role of Sabroxy® in improving glucose tolerance and supporting cognitive function in individuals exhibiting early metabolic and neurocognitive dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male, adults grouped by age as follows 2 groups of 70 patients each (35 active and 35 placebo )

   * GROUP 1 = aged 40 - 60, and
   * GROUP 2 = aged 61 - 80
2. In good general health
3. Screening HOMA-IR value ≥ 2.0 to < 4.0
4. Screening fasting glucose 100 to 135 mg/dL
5. Screening MoCA less than 26

Exclusion Criteria:

1. Having been diagnosed with known allergies to any ingredients in the study product.
2. Relevant history or presence of any medical disorder potentially interfering with this study (e.g., malabsorption, chronic gastrointestinal diseases, severe depression, cardiovascular disease occurrence within the last 3 months, etc.),
3. Regular intake of medications or supplements known to affect glucose tolerance
4. Breastfeeding, pregnant, or planning to become pregnant during the study, according to the subject's self-report.
5. Having a pregnant partner or a partner who is planning to become pregnant during the study period or is unwilling or unable to use an acceptable method of contraception.
6. Having a history of skin cancer within the past 5 years.
7. Having a history of immunosuppression/immune deficiency disorders (including HIV infection, it has been AIDS, multiple sclerosis, Crohn's disease, rheumatoid arthritis), organ transplant (heart, kidney, etc.), or currently using oral or systemic immunosuppressive medications and biologics (e.g., azathioprine, belimumab, Cimzia®, Cosentyx®, cyclophosphamide, cyclosporine, Enbrel®, Humira®, Imuran®, Kineret®, mycophenolate mofetil, methotrexate, Orencia®, prednisone, Remicade®, Rituxan®, Siliq™, Simponi®, Stelara®, Taltz®) and/or undergoing radiation or chemotherapy as determined by study documentation.
8. Currently using or having regularly used corticosteroids (systemic or topical, not nasal or ocular) within the past 4 weeks (including but not limited to betamethasone, clobetasol, desoximetasone, diflorasone, fluocinonide, halcinonide, and halobetasol).
9. Having a disease such as asthma, diabetes, epilepsy, hypertension, hyperthyroidism, or hypothyroidism that is not controlled by diet or medication. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
10. Having started a long-term medication within the last 2 months.
11. Having planned surgeries or invasive medical procedures during the study. Non-invasive medical procedures or surgeries will be reviewed for their impact on the study outcome and acceptability by the Investigator or designee.
12. Currently participating in any other clinical trial at SFRI or another research facility or doctor's office.
13. Having participated in any other clinical trial that evaluates or applies interventions to the same body system, organ, or condition being studied in this trial within 12 weeks prior to the screening visit at SFRI or another research facility or doctor's office.
14. Note - Medications for treatment of chronic diseases that do not affect the metabolism of the study product will be permitted and will be judged individually regarding interference with the study by an investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Resistance as Assessed by HOMA-IR | Prescreening -14 days and Week 8
  Insulin resistance will be evaluated using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting glucose and fasting insulin levels.
  The objective is to determine the mean change in HOMA-IR from baseline to Week 8 between the Sabroxy® and placebo groups.

SECONDARY OUTCOMES:
Change in Cognitive Function Scores (Immediate Word Recall Test) | Baseline- Day 1 and Week 8
  Cognitive performance will be assessed using the Immediate Word Recall test to evaluate short-term memory and verbal learning. The mean change in recall score from baseline to Week 8 will be compared between groups.
Change in Working Memory Performance (Numeric Working Memory Test) | Baseline- Day 1 and Week 8
  Numeric Working Memory test will assess attention, working memory capacity, and processing speed. The change in mean score from baseline to Week 8 will be evaluated between Sabroxy® and placebo groups.
Change in Self-Perceived Cognitive Failures (Cognitive Failures Questionnaire-CFQ) | Baseline- Day 1 and Week 8
  Participants' self-reported everyday cognitive lapses will be evaluated using the Cognitive Failures Questionnaire (CFQ), a 25-item self-assessment scale that measures the frequency of attention, perception, memory, and action failures in daily life.
  Each item is scored on a 5-point Likert scale (0 = never, 4 = very often), yielding a total score range of 0 to 100, with higher scores indicating greater perceived cognitive failures (worse performance).
  The change in CFQ total score from baseline to Week 8 will be analyzed to assess improvement in self-perceived cognitive function.
Change in Montreal Cognitive Assessment (MoCA) Total Score | Prescreening -14 days and Week 8
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a 30-point screening tool designed to detect mild cognitive impairment.
  The total score ranges from 0 to 30, with higher scores indicating better global cognitive performance.
  The change in MoCA total score from baseline to Week 8 will be analyzed to evaluate overall cognitive improvement following intervention.
Change in Serum Brain-Derived Neurotrophic Factor (BDNF) | Prescreening -14 days and Week 8
  Serum BDNF levels will be quantified to assess neuroplasticity response. Mean change in BDNF concentration from baseline to Week 8 will be compared between study groups.
Change in Inflammatory Biomarker (High-Sensitivity C-Reactive Protein, hs-CRP) | Prescreening -14 days and Week 8
  Systemic inflammation will be assessed through serum hs-CRP concentration. Mean change from baseline to Week 8 will be compared between Sabroxy® and placebo groups.
Change in Oxidative Stress Biomarkers- Malondialdehyde (MDA) Concentration | Prescreening -14 days and Week 8
  Oxidative stress will be assessed by measuring malondialdehyde (MDA) levels in serum using a validated spectrophotometric assay.
  MDA is a biomarker of lipid peroxidation, and its concentration will be expressed in micromoles per liter (µmol/L).
  The change in MDA concentration from baseline to Week 8 will be analyzed to evaluate the effect of Sabroxy® supplementation on oxidative stress.
Change in Serum Phosphorylated Tau/Amyloid Beta Ratio (p-Tau/Aβ) | Prescreening -14 days and Week 8
  The ratio of phosphorylated tau to amyloid beta will be evaluated as a neurodegeneration-related biomarker. Mean change from baseline to Week 8 will be compared between groups.
Change in Superoxide Dismutase (SOD) Activity | Prescreening -14 days and Week 8
  Antioxidant enzyme activity will be evaluated by measuring superoxide dismutase (SOD) activity in serum using a validated spectrophotometric method.
  SOD activity will be expressed in units per milliliter (U/mL), where higher activity indicates greater antioxidant defense.
  The change in SOD activity from baseline to Week 8 will be analyzed to assess improvements in antioxidant status.
Change in Glutathione Peroxidase (GPx) Activity | Prescreening -14 days and Week 8
  Antioxidant defense will also be evaluated through glutathione peroxidase (GPx) enzyme activity in serum, measured via a validated spectrophotometric assay.
  GPx activity will be expressed in units per milliliter (U/mL), with higher values indicating stronger antioxidant protection.
  The change in GPx activity from baseline to Week 8 will be analyzed to determine the impact of Sabroxy® on enzymatic antioxidant function.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No